CLINICAL TRIAL: NCT01228357
Title: Predict Antidepressant Responsiveness Using Pharmacogenomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Doh Kwan Kim, M.D., Ph.D., Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2003-08-07
Record Dates: First submitted 2010-10-24; First posted 2010-10-26 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Depressive Symptoms
Keywords: Pharmacogenomics; Depressed Patients
MeSH Terms: conditions — Depression | interventions — Paroxetine; Milnacipran; Nortriptyline; Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SSRI treated group (Experimental): SSRI treated group is patients treated with fluoxetine, paroxetine, or sertraline
  Interventions: Drug: SSRI treated group
- non-SSRI treated group (Active Comparator): non-SSRI treated group is patients treated with milnacipran, venlafaxine, nortriptyline, or mirtazapine
  Interventions: Drug: non-SSRI treated group

INTERVENTIONS:
Drug: SSRI treated group — Antidepressant administration of SSRI class for 12 weeks under therapeutic dose
  Other Names: fluoxetine_Prozac; paroxetine_Paxil, Seroxat; sertraline_Zoloft
  Arms: SSRI treated group
Drug: non-SSRI treated group — Antidepressant administration of non-SSRI class for 12 weeks under therapeutic dose
  Other Names: milnacipran; venlafaxine_Effexor; nortriptyline_Aventyl, Pamelor, Noritren; mirtazapine_Avanza, Zispin, Remeron
  Arms: non-SSRI treated group

SUMMARY:
The purpose of this study is to determine whether genetic information associated with individual depressive symptoms.

DETAILED DESCRIPTION:
The primary hypothesis is that the variations of the candidate genes are associated with individual symptoms in patients with depression.

The Second hypothesis is that patients with the associated genetic variation suffer longer from the associated symptom than the patients without the associated genetic variation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were enrolled in the clinical trials program of hte Samsung Medical Center Geropsychiatry and Affective Disorder Clinics(Seoul, Korea). They received a semistructured diagnostic interview, the Samsung Psychiatric Evaluation Schedule. The affective disorder section of the Samsung Psychiatric Evaluation Schedule uses the Korean version of the structured clinical interview for the diagnostic and statistical manual of mental disorders, Fourth edition.
* interview with one more patient's family member for objective diagnosis and final diagnosis decision by agreements of two more psychiatric physicians

Exclusion Criteria:

* received psychotropic medication within 2 weeks of the study or fluoxetine within 4 weeks
* potential study participants for pregnancy, significant medical conditions, abnormal laboratory baseline values, unstable psychiatric features(eg.suicidal), history of alcohol of drug dependence, seizures, head trauma with loss of consciousness, neurological illness, or concomitant Axis I psychiatric disorder.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2003-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Presences of each individual symptom of depression at 1,2,4,6,12 weeks | 12 weeks
  17-items HAM-D scale was employed to measure depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Kangnam, Seoul, South Korea